CLINICAL TRIAL: NCT06603987
Title: Phase I/II Basket Trial: Boron Neutron Capture Therapy (BNCT) Using CICS-1 and SPM-011 for Patients With Recurrent Solid Malignant Thoracic Tumors That Are Unresectable and Perceived Challenging to Treat With Standard Treatment
Brief Title: Using CICS-1 and SPM-011 and ［18F］FBPA Commissioned by CICS and Sumitomo Heavy Industries and STELLA PHARMA
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stella Pharma Corporation (Industry)
Collaborators: Cancer Intelligence Care Systems, Inc. (Industry); Sumitomo Heavy Industries, Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJ-BT001
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Thoracic Solid Malignant Tumor
Keywords: Esophageal Cancer; Non Small Cell Lung Cancer; Breast Cancer; Malignant Soft Tissue Sarcoma; Malignant Pleural Mesothelioma; Malignant Peripheral Nerve Sheath Tumors
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Mesothelioma, Malignant; Neurofibrosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Boron Neutron Capture Therapy (BNCT) (Experimental)
  Interventions: Radiation: BNCT; Diagnostic Test: ［18F］FBPA

INTERVENTIONS:
Radiation: BNCT — Patients will be infused SPM-011 intravenously at a dose of 200mg/kg/hr over 2 hours. Thereafter, patient will be infused SPM-011 intravenously at a dose of 100mg/kg/hr and will receive neutron irradiation simultaneously for a certain period of time based on his Boronophenylalanine (BPA) concentration in the blood.
Diagnostic Test: ［18F］FBPA — Intravenous injection of ［18F］FBPA and radiation exposure from PET-CT scan.

SUMMARY:
To evaluate the safety and efficacy of Boron Neutron Capture Therapy (BNCT) in patients with recurrent thoracic solid tumors that are difficult to treat with standard radiation therapy or drug therapy and are unresectable. With "lung," "heart," "liver," "spinal cord," and "esophagus" as common risk organs in the treatment plan for BNCT using therapeutic CT to evaluate the safety and efficacy of BNCT in patients with unresectable and recurrent thoracic solid tumors which are difficult to treat with standard radiation and drug therapy.

To evaluate the safety of ［18F］FBPA synthesized with MPS200FBPA. In addition, the usefulness of ［18F］FBPA-PET testing to determine the appropriateness of performing BNCT will be evaluated in an exploratory manner.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained from the subject.
* Patients with histopathological diagnosed malignant tumor (except cutaneous angiosarcoma)
* Measurable disease, as defined by RECIST v1.1.
* Patients diagnosed with recurrent malignant tumors that are unresectable and perceived challenging to treat with standard treatment.
* Patients with ECOG performance status score of 0 or 1.

Exclusion Criteria:

* Patients with active disease or active double cancers other than target lesions.
* Patients with imaging findings that affect imaging evaluation of the tumor, such as ground-glass opacities
* Patients who received radiation therapy exceeding 65 Gy as a prior treatment for the target lesion.
* Any serious concomitant disease that precludes completion of the study treatment.
* Patients with remaining complications of Grade 3 or higher related to prior radiation therapy in the irradiation field.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence rate of dose-limiting toxicity | Baseline until Day180
RECIST v1.1 | Baseline until Day180

CONTACTS AND LOCATIONS:
Locations (1):
- ORIX Kouraibashi Bldg. 8F 3-2-7 Kouraibashi Chuo-ku, Osaka, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No